CLINICAL TRIAL: NCT01971853
Title: Does Preventive Analgesia Improve the Outcome of Demerol-Vistaril Procedural Sedations in Pediatric Dentistry?
Brief Title: Does Preventive Analgesia Improve the Outcome of Demerol-Vistaril Procedural Sedations in Pediatric Dentistry
Acronym: Analgesia
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient number of participants recruited
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 13-1753
Record Dates: First submitted 2013-10-18; First posted 2013-10-29 (Estimated); Results first posted 2021-01-22 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2020-12

CONDITIONS: Pain
Keywords: Analgesia
MeSH Terms: conditions — Pain; Agnosia | interventions — Analgesics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- oral placebo (Placebo Comparator): an Ibuprofen and Acetaminophen Placebo will be added to a Demerol-Vistaril regimen
  Interventions: Drug: oral placebo
- Oral Analgesics (Active Comparator): 5 mg/kg ibuprofen + 15 mg/kg acetaminophen will be added to a Demerol-Vistaril regimen
  Interventions: Drug: Oral Analgesics

INTERVENTIONS:
Drug: oral placebo — Ibuprofen placebo and Acetaminophen placebo will be added to a Demerol-Vistaril regimen
  Other Names: Flavored liquid
  Arms: oral placebo
Drug: Oral Analgesics — Ibuprofen at 5.0 mg/kg and Acetaminophen at 15.0 mg/kg will be added to a Demerol-Vistaril regimen
  Arms: Oral Analgesics

SUMMARY:
All healthcare providers strive continually to improve the outcome of their treatment approaches. The investigators hypothesize that preventive analgesics administered before a child is sedated with a Demerol-Vistaril regimen will improve the outcome of a sedation.

DETAILED DESCRIPTION:
To increase outcomes for patients receiving dental sedation by providing significant evidence that the new regimen improves the quality of sedation and results in an improved post sedation ability to eat, drink, resume normal activities and require less additional pain medications.

ELIGIBILITY:
Inclusion Criteria:

* We intend to enroll 300 children between the ages of 2 - 8 years of all ethnicities for this prospective, placebo controlled, randomized, and double-blind trial. All children that fulfill our general selection criteria for this sedation regimen will be eligible for this study.

Exclusion Criteria:

* Children who do not meet our general selection criteria for this sedation regimen will be ineligible for this study.

Ages: 2 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 88 (Actual)
Dates: Start 2013-10; Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey O Young, DDS, Study Director — University of Colorado, Denver
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study was terminated and the PI has left the institution. Significant efforts were made to obtain the data by contacting the PI/study team members, but those efforts were unsuccessful. No study data are available.
Period: Overall Study
Arm/Group | Oral Placebo | Oral Analgesics
Started | 0 | 0
Completed | 0 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The study was terminated and the PI has left the institution. Significant efforts were made to obtain the data by contacting the PI/study team members, but those efforts were unsuccessful. No study data are available.
Groups:
- Total: Total of all reporting groups
Arm/Group | Oral Placebo | Oral Analgesics | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical
Age, Continuous
Sex: Female, Male
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Improved Sedation Effectiveness Based on Numerical Value for Effectiveness as Noted in Description
Description: A Sedation effectiveness evaluation criteria chart will be utilized to determine a numerical value for the effectiveness as follows:
  1 = Effective/Excellent; 2 = Partially effective/good; 3 = Ineffective/fair; 4 = Aborted/Poor
Time Frame: 60 minutes treatment started
Population: as for baseline characteristics
Arm/Group | Oral Placebo | Oral Analgesics
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Difference in Heart Rate as Measured by Numerical Delta Value
Description: A baseline heart rate will be determined at the beginning of the appointment, and a maximum heart rate will be determined during the appointment. The differences between baseline and maximum heart rates for each study arm will be compared.
Time Frame: From state of treatment (time 0) 60 minutes
Population: as for baseline characteristics
Arm/Group | Oral Placebo | Oral Analgesics
Number analyzed (Participants) | 0 | 0

3. Other Pre Specified Outcome: Time of Administration of Nitrous Oxide and Oxygen as Measured by Minutes and Percent of Nitrous Oxide Administered
Description: The differences in time and concentration of nitrous oxide used during treatment will be compared for each study arm.
Time Frame: From start of treatment (time 0) to 60 minutes
Population: as for baseline characteristics
Arm/Group | Oral Placebo | Oral Analgesics
Number analyzed (Participants) | 0 | 0

4. Other Pre Specified Outcome: Complexity of Procedures Completed as Measured by Numerical Value Using Procedure Complexity Scale in Description
Description: A table will be used to determine the complexity of procedures performed by assigning a numerical value to each procedure and determining a total procedure complexity score.
Time Frame: 60 minutes after start of treatment
Population: as for baseline characteristics
Arm/Group | Oral Placebo | Oral Analgesics
Number analyzed (Participants) | 0 | 0

5. Other Pre Specified Outcome: Complications During Treatment and Recovery
Description: The occurrence of Complications during treatment and recovery will be evaluated. Complications are defined as vomiting, excessive crying, need for supplemental oxygen, and disorientation.
Time Frame: 2 hours in clinic
Population: as for baseline characteristics
Arm/Group | Oral Placebo | Oral Analgesics
Number analyzed (Participants) | 0 | 0

6. Other Pre Specified Outcome: Post Operative Problems
Description: Presence of Post op problems including time and whether problem is constant or intermittent will be as follows: Discomfort when eating/drinking (D), Resumption of normal activity (NA), and Need for additional pain meds (PM)
Time Frame: 4 hours after patient is discharged
Population: as for baseline characteristics
Arm/Group | Oral Placebo | Oral Analgesics
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: The study was terminated and the PI has left the institution. Significant efforts were made to obtain the data by contacting the PI/study team members, but those efforts were unsuccessful. No study data are available.
Arm/Group | Oral Placebo | Oral Analgesics
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
The study was terminated early due to recruitment issues. The PI has left the institution. Significant efforts were made to obtain the data by contacting the PI and the study team members, but those efforts were unsuccessful and we could obtain no results data. No study data are available.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes